CLINICAL TRIAL: NCT06645054
Title: Smart Hallway for Gait Assessment
Brief Title: Usability of the Smart Hallway System in Clinical Setting
Acronym: SmartHallway
Status: Recruiting | Type: Observational
Sponsor: University Rehabilitation Institute, Republic of Slovenia (Other)
Responsible Party: Sponsor
Other Study IDs: URIS202404
Record Dates: First submitted 2024-10-11; First posted 2024-10-16 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Amputation; Gait Disorders, Neurologic
Keywords: Gait analysis; Computerised assessment; Rehabilitation; Lower limb loss; Prosthetics and orthotics
MeSH Terms: conditions — Gait Disorders, Neurologic | interventions — Artificial Limbs

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- LLL: Rehabilitation patients with lower limb loss
  Interventions: Behavioral: Standard rehabilitation; Device: Lower-limb prosthesis
- LLO: Rehabilitation patients fitted with a lower limb orthosis
  Interventions: Behavioral: Standard rehabilitation; Device: Lower-limb orthosis

INTERVENTIONS:
Behavioral: Standard rehabilitation — The patients will receive standard rehabilitation that comprises assessment performed by a multidisciplinary team (physical-and-rehabilitation-medicine specialist physician, physiotherapist, occupational therapist, psychologist, social worker, prosthetics-and-orthotics engineer).
Device: Lower-limb prosthesis — The patients from the LLL group will be fitted with an appropriate lower-limb prosthesis.
  Groups: LLL
Device: Lower-limb orthosis — The patients from the LLO group will be fitted with an appropriate lower-limb orthosis.
  Groups: LLO

SUMMARY:
The aim of the study is to examine suitability of data and processed reports acquired from the Smart Hallway system for clinical settings in terms of user acceptability and accuracy for use in clinical practice.

DETAILED DESCRIPTION:
The goal of the study is to use off-the-shelves markerless and contactless technologies and automatically digitise the person's movements as they walk through an institutional hallway. Multi-camera-based technologies can merge 2D-video into 3D-information. With an appropriate software, one can acquire data, perform the kinematic calculations and generate a report, all with minimal or no human intervention. The specific research question are whether pathological gait or walking disorders of the patients can be identified and classified based on the system's output, whether signs of depression can be classified from the the system's output, and whether the results of the 6-minute walk test can be predicted from the the system's output.

ELIGIBILITY:
Inclusion Criteria:

* ability to walk at least 10 metres without help of a person,
* no severe cognitive problems (able to answer questionnaires),
* native Slovenian speakers,
* wiling to participate (signed informed consent)

Exclusion Criteria:

* severe cognitive impairment,
* not being able to walk with or without a prosthesis or orthosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients after lower limb loss (because of traumatic reason or disease) for the LLL group; patients fitted with lower-limb orthosis because of neurological reasons for the LLO group
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-03-24 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Smart Hallway | Upon admission to rehabilitation
  As part of the regular clinical examination, the patients walk straight through a 7m long walkway, turn, and come back while data is collected with the Smart Hallway system. They start walking one meter outside the capture volume. The procedure is repeated five times to provide a sufficient number of walking cycles. Three-dimensional temporospatial gait features (position, joint angles, velocities, accelerations) are extracted from the acquired data.
Falls during rehabilitation | Upon discharge from rehabilitation
  Data on falls during rehabilitation is routinely collected and entered in the hospital information system (HIS). It will be transferred from the HIS to the study database upon the patient's discharge.

SECONDARY OUTCOMES:
World Health Organisation Disability Assessment Schedule | Upon admission to rehabilitation
  The World Health Organisation Disability Assessment Schedule (WHODAS II) is a generic patient-reported outcome measure of disability that has been translated into Slovenian. It covers six life domains. The scores range from 0 to 100; higher score indicates more disability (i.e., worse outcome).
Activity Specific Balance Confidence Scale | Upon admission to rehabilitation
  The Activity Specific Balance Confidence Scale (ABC) is a pathology-specific patient-reported outcome measure of balance that has been translated and validated in Slovenian. The scores range from 0 to 100; higher score indicates more confidence (i.e., better outcome).
Hospital Anxiety and Depression Scale | Upon admission to rehabilitation
  The Hospital Anxiety and Depression Scale (HADS) is a patient-reported outcome measure that is used for assessing depression, which has been translated and validated in Slovenian. The scales comprises 14 items, 7 for anxiety and 7 for depression, all scored from 0 to 3, so the score range is from 0 to 21 for either anxiety or depression. Higher score means more pronounced anxiety and depression (i.e., worse outcome).
Six-minute walk test | Upon admission to rehabilitation
  The Six-minute Walk Test (6MWT) is a standard test for assessing walking speed over a long distance with good and well-known metric characteristics. Longer walked distance means higher walking speed (i.e., better outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Helena Burger, MD, PhD, Principal Investigator — University Rehabilitation Institute, Republic of Slovenia
Locations (1):
- University Rehabilitation Institute, Republic of Slovenia, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Undecided